CLINICAL TRIAL: NCT02605265
Title: A Randomized Phase III Trial of Capecitabine With or Without Irinotecan Driven by UGT1A1 in Neoadjuvant Chemoradiation of Locally Advanced Rectal Cancer
Brief Title: Trial of Capecitabine With or Without Irinotecan Driven by UGT1A1
Acronym: CinClare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Hubei Cancer Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-R005
Record Dates: First submitted 2015-11-09; First posted 2015-11-16 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Neoadjuvant Chemoradiation; Irinotecan; UGT1A1
MeSH Terms: interventions — Radiation; Capecitabine; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine Alone (Active Comparator): Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 825mg/m2 bid Monday-Friday per week
  Chemotherapy in Interval Between CRT and Surgery:
  Capecitabine: 1000mg/m2 bid d1-14; Oxaliplatin: 130mg/m2 d1
  Surgery:
  Scheduled 6-8 weeks after the completion of CRT
  Adjuvant Chemotherapy:
  Capecitabine: 1000mg/m2 bid d1-14; Oxaliplatin: 130mg/m2 d1; q3w, 5cycles
  Interventions: Radiation: Radiation; Drug: Capecitabine; Drug: Oxaliplatin
- Capecitabine with Irinotecan (Experimental): Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7)
  Chemotherapy in Interval Between CRT and Surgery:
  Capecitabine: 1000mg/m2 bid d1-14; Irinotecan: 200mg/m2 d1
  Surgery:
  Scheduled 6-8 weeks after the completion of CRT
  Adjuvant Chemotherapy:
  Capecitabine: 1000mg/m2 bid d1-14; Oxaliplatin: 130mg/m2 d1; q3w, 5cycles
  Interventions: Radiation: Radiation; Drug: Capecitabine; Drug: Irinotecan; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: Radiation — Pelvic Radiation: 50Gy/25Fx
Drug: Capecitabine
  Other Names: Xeloda
Drug: Irinotecan
  Other Names: CPT-11
  Arms: Capecitabine with Irinotecan
Drug: Oxaliplatin

SUMMARY:
The study evaluate the addition of Irinotecan in neoadjuvant chemoradiation. Half of participants will receive capecitabine alone together with neoadjuvant CRT, followed by a cycle of XELOX, while the other will receive capecitabine and irinotecan during CRT, followed by a cycle of XELIRI. All participants will be scheduled to receive surgery 6-8 weeks after the completion of CRT, then 5 cycles of adjuvant chemotherapy of XELOX.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed adenocarcinoma
* clinical stage T3-4 and/or N+
* the distance from anal verge less than 12 cm
* without distance metastases
* KPS >=70
* UGT1A1*28 6/6 or 6/7
* without previous anti-cancer therapy
* sign the inform consent

Exclusion Criteria:

* pregnancy or breast-feeding women
* serious medical illness
* baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
* DPD deficiency
* UGT1A1*28 7/7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response | Surgery scheduled 6-8 weeks after the end of chemoradiation

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 10 years
Disease-free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 years
Local Control rate | From date of randomization until the date of first documented pelvic failure, assessed up to 10 years
  Number of participants with pelvic failure after surgery, evaluated using Kaplan-Meier Curve
Number of participants with chemoradiation-related adverse events as assessed by CTCAE v4.0 | Up to 2 years
Surgical complications | Surgery scheduled 6-8 weeks after the end of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Z, Sun X, Liu A, Zhu Y, Zhang T, Liu L, Jia J, Tan S, Wu J, Wang X, Zhou J, Yang J, Zhang C, Zhang H, He X, Cai G, Huang C, Xia F, Wan J, Zhang H, Shen L, Wang L, Zhang W, Cai S, Zhu J. Neoadjuvant chemoradiotherapy with capecitabine and irinotecan guided by UGT1A1 status in patients with locally advanced rectal cancer: 5-year update of the CinClare trial. Cancer Commun (Lond). 2025 Nov;45(11):1417-1430. doi: 10.1002/cac2.70058. Epub 2025 Sep 3. PMID 40899645
- [Derived] Zhang X, Fan J, Zhang L, Wang J, Wang M, Zhu J. Association Between Three-Dimensional Transrectal Ultrasound Findings and Tumor Response to Neoadjuvant Chemoradiotherapy in Locally Advanced Rectal Cancer: An Observational Study. Front Oncol. 2021 Jun 4;11:648839. doi: 10.3389/fonc.2021.648839. eCollection 2021. PMID 34178635
- [Derived] Zhu J, Liu A, Sun X, Liu L, Zhu Y, Zhang T, Jia J, Tan S, Wu J, Wang X, Zhou J, Yang J, Zhang C, Zhang H, Zhao Y, Cai G, Zhang W, Xia F, Wan J, Zhang H, Shen L, Cai S, Zhang Z. Multicenter, Randomized, Phase III Trial of Neoadjuvant Chemoradiation With Capecitabine and Irinotecan Guided by UGT1A1 Status in Patients With Locally Advanced Rectal Cancer. J Clin Oncol. 2020 Dec 20;38(36):4231-4239. doi: 10.1200/JCO.20.01932. Epub 2020 Oct 29. PMID 33119477
- [Derived] Yao Y, Xu X, Yang L, Zhu J, Wan J, Shen L, Xia F, Fu G, Deng Y, Pan M, Guo Q, Gao X, Li Y, Rao X, Zhou Y, Liang L, Wang Y, Zhang J, Zhang H, Li G, Zhang L, Peng J, Cai S, Hu C, Gao J, Clevers H, Zhang Z, Hua G. Patient-Derived Organoids Predict Chemoradiation Responses of Locally Advanced Rectal Cancer. Cell Stem Cell. 2020 Jan 2;26(1):17-26.e6. doi: 10.1016/j.stem.2019.10.010. Epub 2019 Nov 21. PMID 31761724
- [Derived] Guan Y, Shen Y, Xu Y, Li C, Wang J, Gu W, Lian P, Huang D, Cai S, Zhang Z, Zhu J. An expansion study of genotype-driven weekly irinotecan and capecitabine in combination with neoadjuvant radiotherapy for locally advanced rectal cancer with UGT1A1 *1*1 genotype. Therap Adv Gastroenterol. 2019 Jun 6;12:1756284819852293. doi: 10.1177/1756284819852293. eCollection 2019. PMID 31217818